CLINICAL TRIAL: NCT05849831
Title: The Role of Ultrasonographic Assessment of Optic Nerve Sheath Diameter in Prediction of Sepsis Associated Encephalopathy
Brief Title: Optic Nerve Sheath Diameter for Prediction of Sepsis Associated Encephalopathy
Status: Completed | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Sherif M. S. Mowafy, associate professor of anaesthesia and intensive care, Zagazig University
Other Study IDs: 10597-30-4-2023
Record Dates: First submitted 2023-02-11; First posted 2023-05-09 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult critically ill septic patients
  Interventions: Diagnostic Test: Ultrasound measurement of Optic nerve sheath diameter

INTERVENTIONS:
Diagnostic Test: Ultrasound measurement of Optic nerve sheath diameter — Ocular ultrasonography will be performed by single skilled examiner with patients placed in supine position with closed eyes. A layer of ultrasound gel will be applied over the closed upper eyelid and the liner high frequency probe 7 - 12 MHz of SonoSite M-Turbo ultrasound machine is placed on temporal area of eyelid with the hand holding it resting on forehead of patient. ONSD is measured 3mm behind the globe in the transverse plane perpendicular to the optic nerve. For each eye one measurement will be made and the reported ONSD corresponds to the mean of the two values obtained for each patient. An average ONSD greater than 5 mm is considered abnormal and elevated intracranial pressure should be suspected. all enrolled subjects will be eligible for ONSD measurements, SOFA score calculation, as well as GCS assessment on daily basis for up to 10 consecutive days, until ICU discharge or death.

SUMMARY:
Sepsis-associated brain dysfunction (SABD)with increased intracranial pressure is a complex pathology that can lead to unfavourable outcome. Although direct measurement of intracranial pressure using an intra-ventricular catheter remains the gold standard, it is burdened with potential serious complications due to its invasiveness. Ultrasonic measurement of optic nerve sheath diameter (ONSD) is a non-invasive method for ICP monitoring.

Screening for SABD is crucial for early diagnosis and management, measurement of ONSD can detect elevated intracranial pressure in septic patients. Intracranial hypertension in septic patients might be a sign of SABD.

Using ONSD for SABD screening requires further research. So, we hypothesized that ONSD could be used as an objective screening tool to predict and early diagnose SABD in adult septic patients.

DETAILED DESCRIPTION:
Sepsis is the most common complication in adult critically ill patients, and it has been become the leading cause of morbidity and mortality worldwide. The essential component of sepsis is the presence of an acute organ dysfunction. The brain is highly vulnerable to the inflammatory storm associated with infection and it may be the first organ to show signs of life-threatening organ dysfunction caused by infection. This brain dysfunction is known as "sepsis-associated encephalopathy (SAE)".

Sepsis-associated brain dysfunction is considered the commonest type of encephalopathy seen in intensive care unit (ICU). it is defined as a life- threatening acute diffuse brain dysfunction due to infection outside the central nervous system (CNS) and is mostly caused by the inflammatory storm. It varies from delirium or confusion, seizure or focal neurological sign, and diffuse or multifocal neurological deficits, to stupor or coma with no other diagnoses describing the patient neurological status. SAE may occur in up to 70% of septic patients and it significantly increases mortality. It is a complex syndrome with unclear pathophysiology. The possible causes could include neuro-inflammation, excitotoxicity, impaired cerebral autoregulation, and cerebral ischemia. These Pathophysiological changes may lead to increase in the intracranial pressure (ICP) which may in turn decrease cerebral perfusion and lead to brain edema, brain damage and compromised the outcome of these patients. Therefore, early detection of increased ICP is of paramount importance for timely intervention and improved prognosis. However, direct invasive ICP monitoring is not routinely recommended in non-traumatic coma patients as well as septic patients either due to absence of intracranial infection or coagulopathy; so, a reliable non-invasive ICP monitoring method is highly recommended. Bedside ultrasonographic assessment of the optic nerve sheath diameter (ONSD) offers a satisfactory non-invasive ICP monitoring test and is documented as a sensitive and specific predictor of cerebral edema and is strongly correlated with both invasive ICP measurements and radiographic cerebral edema as diagnosed by CT scan or MRI.

Considering that SAE is a diagnosis of exclusion as well as screening method for SAE is necessary for early diagnosis and timely management. We hypothesized that ONSD could have a role as an objective screening tool to predict and early diagnose ICP changes in septic patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient acceptance.
* Age 21- 70 years old.
* Patients diagnosed with sepsis For diagnosis of sepsis and septic shock, the third international definition and appropriate diagnostic criteria was used.

Sepsis was defined as life-threatening organ dysfunction caused by a dysregulated host response to an infection, and it is suspected in an acutely deteriorating patient in whom there is clinical evidence or strong suspicion of infection. Septic shock was defined as the need for vasopressors or vasoactive medication to maintain a mean arterial blood pressure of 65 mmHg or higher after adequate fluid resuscitation, with the presence of a high lactate (>2 mmol/l).

Exclusion Criteria:

* Patient refusal.
* Ocular wound
* History of prior ocular trauma or surgery
* Conjunctival edema or orbital edema
* Vitreous hemorrhage
* Central nervous system (CNS) infection
* Cerebrovascular accident
* Brain trauma
* Any previous neurosurgical procedure

Ages: 21 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with sepsis will be enrolled and the severity of clinical illness will be assessed using APACHE II on ICU admission. SOFA will be calculated daily.
  Patients who have changes in mental state, especially in consciousness and cognition, and other factors that cause mental changes were excluded as well as brain CT already ordered. Therefore, managing ICU team decided to diagnose patient with SAE.
  Accordingly, patients will be divided into non-SAE group: include fully conscious patients suffering from sepsis for fewer than 24 h.
  SAE group: include patients with sepsis for fewer than 24 h, suffering from acute onset of disturbed conscious level.
  All enrolled subjects will undergo ONSD assessment within 24 h of admission and they will be eligible for ONSD measurements, SOFA score calculation, as well as GCS assessment on daily basis for up to 10 consecutive days, until ICU discharge or death.
Sampling Method: Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2023-05-03 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
correlation between ONSD measurements and the occurrence of SAE | 10 days
  ultrasonographic measurement of optic nerve sheath diameter (ONSD) will be performed and recorded on daily basis for up to 10 consecutive days, until ICU discharge or death then we will compare the ONSD measurements of non-SAE patients to those of SAE patients.

SECONDARY OUTCOMES:
the correlation between ONSD measurements and the ICU mortality of critically ill patients with sepsis | 30 days
  ultrasonographic measurement of optic nerve sheath diameter (ONSD) will be performed and recorded on daily basis for up to 10 consecutive days, until ICU discharge or death then we will compare the ONSD measurements of ICU survivors to those of dead patients during the ICU stay.

CONTACTS AND LOCATIONS:
Overall Officials: Sherif MS Mowafy, MD, Principal Investigator — Anaesthesia, Intensive Care, and Pain Management Department. Faculty of Medicine, Zagazig University,
Locations (2):
- Egypt (2):
  - Benha University Hospitals, Banhā, Qalyubia Governorate
  - Zagazig University Hospitals, Zagazig, Sharqia Province

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: the IPD and any additional supporting information will become available starting 6 months after publication
Access Criteria: by contacting the study investigator

REFERENCES:
- [Background] Coopersmith CM, De Backer D, Deutschman CS, Ferrer R, Lat I, Machado FR, Martin GS, Martin-Loeches I, Nunnally ME, Antonelli M, Evans LE, Hellman J, Jog S, Kesecioglu J, Levy MM, Rhodes A. Surviving sepsis campaign: research priorities for sepsis and septic shock. Intensive Care Med. 2018 Sep;44(9):1400-1426. doi: 10.1007/s00134-018-5175-z. Epub 2018 Jul 3. PMID 29971592
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] 3. Tong D, Wang S, Wang Y, et al. Sepsis-associated Encephalopathy In ICU Admissions: Prevalence, Early Risk of Death, and its Early Prevent and Control. Research Square; 2020. DOI: 10.21203/rs.3.rs-58687/v1.
- [Background] Czempik PF, Pluta MP, Krzych LJ. Sepsis-Associated Brain Dysfunction: A Review of Current Literature. Int J Environ Res Public Health. 2020 Aug 12;17(16):5852. doi: 10.3390/ijerph17165852. PMID 32806705
- [Background] Heming N, Mazeraud A, Verdonk F, Bozza FA, Chretien F, Sharshar T. Neuroanatomy of sepsis-associated encephalopathy. Crit Care. 2017 Mar 21;21(1):65. doi: 10.1186/s13054-017-1643-z. PMID 28320461
- [Background] Crippa IA, Subira C, Vincent JL, Fernandez RF, Hernandez SC, Cavicchi FZ, Creteur J, Taccone FS. Impaired cerebral autoregulation is associated with brain dysfunction in patients with sepsis. Crit Care. 2018 Dec 4;22(1):327. doi: 10.1186/s13054-018-2258-8. PMID 30514349
- [Background] Pfister D, Siegemund M, Dell-Kuster S, Smielewski P, Ruegg S, Strebel SP, Marsch SC, Pargger H, Steiner LA. Cerebral perfusion in sepsis-associated delirium. Crit Care. 2008;12(3):R63. doi: 10.1186/cc6891. Epub 2008 May 5. PMID 18457586
- [Background] Pfister D, Schmidt B, Smielewski P, Siegemund M, Strebel SP, Ruegg S, Marsch SC, Pargger H, Steiner LA. Intracranial pressure in patients with sepsis. Acta Neurochir Suppl. 2008;102:71-5. doi: 10.1007/978-3-211-85578-2_14. PMID 19388291
- [Background] Czempik PF, Gasiorek J, Bak A, Krzych LJ. Ultrasonic Assessment of Optic Nerve Sheath Diameter in Patients at Risk of Sepsis-Associated Brain Dysfunction: A Preliminary Report. Int J Environ Res Public Health. 2020 May 22;17(10):3656. doi: 10.3390/ijerph17103656. PMID 32456003
- [Background] Yang Z, Qin C, Zhang S, Liu S, Sun T. Bedside ultrasound measurement of optic nerve sheath diameter in patients with sepsis: a prospective observational study. Crit Care. 2020 May 18;24(1):235. doi: 10.1186/s13054-020-02959-7. No abstract available. PMID 32423483
- [Background] Cammarata G, Ristagno G, Cammarata A, Mannanici G, Denaro C, Gullo A. Ocular ultrasound to detect intracranial hypertension in trauma patients. J Trauma. 2011 Sep;71(3):779-81. doi: 10.1097/TA.0b013e3182220673. PMID 21909008
- [Background] Rajajee V, Vanaman M, Fletcher JJ, Jacobs TL. Optic nerve ultrasound for the detection of raised intracranial pressure. Neurocrit Care. 2011 Dec;15(3):506-15. doi: 10.1007/s12028-011-9606-8. PMID 21769456
- [Background] Strumwasser A, Kwan RO, Yeung L, Miraflor E, Ereso A, Castro-Moure F, Patel A, Sadjadi J, Victorino GP. Sonographic optic nerve sheath diameter as an estimate of intracranial pressure in adult trauma. J Surg Res. 2011 Oct;170(2):265-71. doi: 10.1016/j.jss.2011.03.009. Epub 2011 Apr 1. PMID 21550065
- [Background] Major R, Girling S, Boyle A. Ultrasound measurement of optic nerve sheath diameter in patients with a clinical suspicion of raised intracranial pressure. Emerg Med J. 2011 Aug;28(8):679-81. doi: 10.1136/emj.2009.087353. Epub 2010 Aug 15. PMID 20713366
- [Background] Qayyum H, Ramlakhan S. Can ocular ultrasound predict intracranial hypertension? A pilot diagnostic accuracy evaluation in a UK emergency department. Eur J Emerg Med. 2013 Apr;20(2):91-7. doi: 10.1097/MEJ.0b013e32835105c8. PMID 22327166
- [Background] Shirodkar CG, Rao SM, Mutkule DP, Harde YR, Venkategowda PM, Mahesh MU. Optic nerve sheath diameter as a marker for evaluation and prognostication of intracranial pressure in Indian patients: An observational study. Indian J Crit Care Med. 2014 Nov;18(11):728-34. doi: 10.4103/0972-5229.144015. PMID 25425840
- [Background] Sekhon MS, Griesdale DE, Robba C, McGlashan N, Needham E, Walland K, Shook AC, Smielewski P, Czosnyka M, Gupta AK, Menon DK. Optic nerve sheath diameter on computed tomography is correlated with simultaneously measured intracranial pressure in patients with severe traumatic brain injury. Intensive Care Med. 2014 Sep;40(9):1267-74. doi: 10.1007/s00134-014-3392-7. Epub 2014 Jul 18. PMID 25034476
- [Derived] Mowafy SMS, Bauiomy H, Kohaf NA, Abd Ellatif SE. The Role of Ultrasonographic Assessment of Optic Nerve Sheath Diameter in Prediction of Sepsis-Associated Encephalopathy: Prospective Observational Study. Neurocrit Care. 2025 Aug;43(1):308-317. doi: 10.1007/s12028-024-02187-9. Epub 2025 Jan 15. PMID 39815108